CLINICAL TRIAL: NCT03496428
Title: Customized Impressions in Dental Implants - Soft Tissues Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implantology Institute (Other)
Collaborators: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: II2017-06
Record Dates: First submitted 2018-03-31; First posted 2018-04-12 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-08

CONDITIONS: Soft Tissue
Keywords: intra-oral scanner; customized impression coping; extra-oral scanner; accuracy

STUDY DESIGN:
Intervention Model Description: To describe the soft tissues dimensional changes (based on STL files) occurred between an intra-oral scanner and standartized scan-body and a extra-oral scanner of stone cast poured from silicone impression with a customized impression coping
  12 months after implant placement and simultaneous regeneration with L-PRF and bovine bone graft in the aesthetic zone of atrophic maxillae in full arch implant supported rehabilitations
Masking Description: Altough it is a single arm two different techniques will be used and obtained STL files will be identified as A and B and the outcomes assessor will not be informed which group corresponds to intra-oral scanner and extra-oral scanner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental implant Impression Techniques (Other): Dental implant impressions- Different Techniques An customized impression coping will be created based on the provisional crown emergence profile which will be used to perform a silicone implant impression. A conventional cast will be created based on the silicone impression and an extra-oral scanner reading will be performed with a 3shape D2000.
  An intra-oral scanner (Trios, 3Shape) will be used to scan the entire arch. The STL file created will be compared and tooth positions and soft tissues discrepancies will be determined
  Interventions: Device: Dental implant impressions- Different Techniques

INTERVENTIONS:
Device: Dental implant impressions- Different Techniques — Assessment of soft tissues changes with different techniques

SUMMARY:
Six patients with a single unit implant in the anterior maxilla (from premolar to premolar), after at least 3 months with provisional implant supported restoration will be submitted to definitive implant impressions.

Informed consents and local ethical committee clearance will be obtained. Patients will be submitted to a silicon impression with a customized impression coping from which a conventional cast will be obtained and scanned with D2000 (3Shape) and to an intraoral scan with Trios (3Shape). Standard Tessellation Language (STL) files will be obtained from both procedures and imported to reverse engineering software Geomagic Control X (3D Systems) and the distance between both scans will be calculated in a colored 3D map. From this map, two outcomes will be analyzed: the changes in soft tissues around implants with the two techniques (primary outcome) and the discrepancy between both scans in the teeth adjacent to the implants (secondary outcome).

DETAILED DESCRIPTION:
"Custom-guided" tissue healing with o provisional restoration is the most predictable way to achieve natural anatomically shaped tissue and optimal esthetics. Several authors describe the use of an anatomically contoured provisional restoration to start to guide the soft tissue healing in an ideal, natural morphology that replicates the tooth form. Being that, after shaping the tissue to ideal anatomic form and health the exact duplication of the soft tissue contour should be obtained so that laboratory can duplicate it in the final restoration. Nowadays gold-standard, describes the use of a customized impression coping that replicates the provisional soft tissue contour by the use of and analog-silicone index upon which a gypsum cast is created.

The use of computer-aided design/computer-assisted manufacture (CAD/CAM) technologies to manufacture prosthetic frameworks on dental implants is noticeably increasing. This method requires the use of an STL file which can be acquired intra-orally or extraorally using a stone cast poured from a conventional implant impression using a customized implant impression coping.

Several studies have already described the accuracy of STL data and that evaluating STL models can be done by best fit algorithms in appropriate softwares.

In this pilot study, the investigators aim to evaluate soft tissue profile changes in single unit implants in the aesthetic area using a customized impression coping with conventional methods and the intraoral impression with an intraoral scanner (Trios, 3Shape). Additionally position discrepancies of adjacent teeth between the two techniques will be assessed.

This pilot study will include 6 patients with single unit implant which will be recruited according inclusion criteria and submitted to the two different impression techniques. Conventional stone cast will be scanned with a laboratory scanner D2000 (3Shape) with a described deviation of 5μm. Two STL files will be obtained per patient and by established methods with a reverse engineering software (Geomagic Control X, 3D Systems) discrepancies between them assessed.

Differences in axis (x, y, z) and overall distances will be assessed in the soft tissues (18 points) and in adjacent teeth (26 points) according established methods, per patient. Additionally, 3D colored maps will be produced to ascertain volumetric changes between techniques. T-test and Wilcoxon signed-rank test will be used and the level of statistical significance set at P<0.05. Sample size determination will be performed based on obtained results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single implant with adjacent teeth in the anterior esthetic area (Pre-Molar to Pre-Molar) of the upper arch with provisional implant crown use and indication for rehabilitation for definitive implant supported crown.

Exclusion Criteria:

- Patients without soft tissue contouring or without provisional implant supported use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duarte Marques, DDS, PhD, Principal Investigator — Implantology Institute; João Caramês, DDS, PhD, Study Director — Implantology Institute; Antonio Mata, DDS, PhD, Principal Investigator — Grupo de Investigação em Bioquímica e Biologia Oral
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: be at least 18 years of age; have at least one implant in the anterior maxilla with the indication for rehabilitation with a definitive implant supported crown; have two mesial and two distal adjacent teeth to the implant and be rehabilitated with a provisional implant supported crown for at least 3 months.
Units Other Than Participants: tooth and implant sites
Groups:
- Dental Implant Impression Techniques: Dental implant impressions- Different Techniques An customized impression coping will be created based on the provisional crown emergence profile which will be used to perform a silicone implant impression. A conventional cast will be created based on the silicone impression and an extra-oral scanner reading will be performed with a 3shape D2000.
  An intra-oral scanner (Trios, 3Shape) will be used to scan the entire arch. The STL file created will be compared and tooth positions and soft tissues discrepancies will be determined
  Dental implant impressions- Different Techniques: Assessment of soft tissues changes with different techniques
Period: Overall Study
Arm/Group | Dental Implant Impression Techniques
Started | 6; 412 tooth and implant sites (304 locations distributed for the analyzed teeth 108 locations distributed for the implant spots)
Completed | 6; 412 tooth and implant sites (304 locations distributed for the analyzed teeth 108 locations distributed for the implant spots)
Not Completed | 0; 0 tooth and implant sites

BASELINE CHARACTERISTICS:
Arm/Group | Dental Implant Impression Techniques
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 51 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Changes in Soft Tissues Around Implant
Description: Discrepancies in soft tissues around implants between different techniques, conventional and digital, in a single unit implant impression, measured as root mean square in µm.
Time Frame: Both techniques will be used in the same appointment upon 3 months use of provisional crown
Population: Patients with a single implant in the esthetic anterior maxillar zone in need of a definitive crown.
Measure: Mean (95% Confidence Interval); unit: root mean square in µm
Arm/Group | Dental Implant Impression Techniques
Number analyzed (Participants) | 6
root mean square in µm | 243.89 [209.15 to 278.63]

2. Secondary Outcome: Discrepancy (Trueness) Between STL Files in Teeth Adjacent to Implant
Description: Linear measurements in µm between STL files in teeth adjacent to implant in several pre-defined locations
Time Frame: Both techniques will be used in the same appointment upon 3 months use of provisional crown
Population: Patients in need of a definitive crown in a single implant in the esthetic anterior maxillar zone.
Measure: Mean (95% Confidence Interval); unit: Root mean square in μm
Arm/Group | Dental Implant Impression Techniques
Number analyzed (Participants) | 6
Root mean square in μm | 51.08 [45.68 to 56.47]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dental Implant Impression Techniques
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03496428/Prot_SAP_000.pdf